CLINICAL TRIAL: NCT06056817
Title: Chronic Evaluation of Novel Pacemaker System
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Calyan Technologies (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: CT-05
Record Dates: First submitted 2023-09-21; First posted 2023-09-28 (Actual); Last update posted 2024-08-20 (Actual); Status verified 2023-09

CONDITIONS: Ventricular Pacing With Rate Response; Bradycardia
MeSH Terms: conditions — Bradycardia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Treatment (Experimental): Chronic implantation of the Calyan pacemaker device
  Interventions: Device: Calyan Pacemaker

INTERVENTIONS:
Device: Calyan Pacemaker — The Calyan pacemaker is a device designed for implantation in the chest below the xiphoid process, and includes a FlexArm containing stimulation and sensing electrodes. The Calyan pacemaker is implanted using a set of delivery tools and clipped onto the xiphoid process; the FlexArm electrodes are oriented to make contact with the pericardial surface of the heart. Pacing parameters are adjusted wirelessly with a tablet-based programmer that communicates with the Calyan pacemaker via secure Bluetooth.

SUMMARY:
The primary study objective is to evaluate the feasibility, initial clinical safety and potential effectiveness of the Calyan Pacemaker system.

DETAILED DESCRIPTION:
This is an early feasibility study, designed to evaluate the initial clinical safety, device functionality and stability and potential effectiveness of the Calyan pacemaker. The Calyan device will be implanted, and if acute success criteria are met, chronic pacing will be delivered over a 3-month primary follow-up period, with subsequent extended follow-up of all patients. The data from this study will be used to justify the design of a larger prospective pivotal study that will assess the safety and effectiveness of the Calyan pacemaker device.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 or above
2. Willing and capable of providing informed consent
3. Class I or IIa indication for implantation of a single-chamber ventricular pacemaker, according to ACC/AHA/HRS guidelines
4. A life expectancy of at least one year, and is a suitable candidate based on overall health and well-being

Exclusion Criteria:

1. Patients with complete AV block or other pacemaker-dependent conditions
2. Patients in whom a substernal device implant should be avoided:

   1. Any prior sternotomy;
   2. Any prior medical condition or procedure that leads to adhesions in the anterior mediastinal space;
   3. Any marked sternal abnormality, such as pectus excavatum or pectus carinatum
   4. Prior abdominal surgery in the epigastric region
   5. Planned sternotomy
   6. Prior or planned chest radiotherapy
   7. Hiatal hernia that distorts mediastinal anatomy
   8. Adhesions in the anterior mediastinal space
   9. Severe obesity so that subxiphoid/substernal tunneling cannot be safely performed
3. Patients with severe RV dilation, gross hepatosplenomegaly, or severe obesity such that subxiphoidal/substernal tunneling cannot be safely performed
4. Patients with a class III indication for a permanent pacemaker
5. Patients with decompensated heart failure not due to bradycardia and expected to worsen with chronic RV pacing
6. Patients with an implanted cardiac pacemaker, cardioverter defibrillator, cardiac resynchronization device, or neurostimulator device, or planned implantation of a cardioverter defibrillator, cardiac resynchronization device, or neurostimulator device
7. Patients with a current or planned implantation of a substernal device, or any implanted device that would interfere with the implantation or operation of a substernal device
8. Patients who have previously undergone an open-heart surgical procedure.
9. Patients with an active infection
10. Patient on chronic oral anticoagulation which cannot be temporarily discontinued for surgery
11. Patients with a condition in which pericardial pacing would be difficult or impossible, such as acute pericarditis, chronic pericardial effusion or pericardial thickening or calcification, cardiac tamponade, or chronic restrictive pericarditis
12. Patients who have tested positive for the COVID-19 in the past 3 months, or are currently showing symptoms consistent with COVID-19
13. Women of childbearing potential who are or might be pregnant at the time of the study or breastfeeding
14. Subjects with a life expectancy of less than 12 months
15. Patients who are currently enrolled or planning to participate in any concurrent clinical study with an investigational therapy
16. Patients with decompensated heart failure expected to worsen with chronic RV pacing
17. Patients with COPD with oxygen dependence

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-10-01 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of procedure and device related serious adverse events (SAEs) | 3 months
  Rate of procedure and device related serious adverse events (SAEs) at 3 months post-implant.
Number of patients with successful chronic ventricular pacing | 3 months
  Proportion of patients with successful chronic ventricular pacing, including successful pacemaker implantation and chronic capture of the ventricle, during the 3-month primary follow-up period.

CONTACTS AND LOCATIONS:
Overall Officials: Imad Libbus, PhD, Study Director — Calyan Technologies
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No